CLINICAL TRIAL: NCT06949839
Title: Effectiveness of a Therapeutic Exercise Program Combined With Respiratory Muscle Training in Patients With Subacute Stroke: a Randomized Clinical Trial
Brief Title: Effectiveness of Therapeutic Exercise Combined With Respiratory Muscle Training in Patients With Subacute Stroke
Acronym: REMUST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Lista Paz (Other)
Collaborators: Complexo Hospitalario Universitario de A Coruña (Other); Universidade da Coruña (Other)
Responsible Party: Sponsor-Investigator, Ana Lista Paz, PhD. Permanent Labor Professor of the Faculty of Physiotherapy at the University of Coruña, Universidade da Coruña
Organization: Universidade da Coruña (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REMUST; 2025/061 (Other: Comité de Ética de la Investigación de A Coruña-Ferrol)
Record Dates: First submitted 2025-04-08; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: stroke; exercise therapy; respiratory muscle training; walk test; physical therapy modalities
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups: the intervention group will perform a combined therapeutic exercise and RMT program, while the control group will combine the same therapeutic exercise program and sham RMT. The duration of the intervention (to both groups) will be eight weeks. The therapeutic exercise program will be carried out three days per week at the CHUAC hospital, and the RMT protocol will be carried out at the home of each patient five days per week, with on-site follow-up every 10 days at the CHUAC. Additionally, half of the subjects from the intervention group will continue the RMT protocol once the eight-week period has ended, with a frequency of two days per week and until the six-month follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, regardless of their group, will perform the same therapeutic exercise program. In addition, they will not know whether their RMT device is sham or not (they have the same appearance). One researcher (physical therapist) will perform both the outcomes assessment and the therapeutic exercise intervention and will be blinded to the group assignment of the patients to the intervention group or the control group. Another researcher (speech therapist) will be responsible for delivering the RMT and sham RMT devices based on the randomization and instructing the patients in their use, as well as increasing the resistance of the valve and re-evaluating the execution of the protocol to confirm that it is being carried out correctly. Therefore, this last therapist will be the only one who will know the group assignments. Mechanisms will be applied to verify whether the masking of both the physiotherapist and the patients to the groups has been violated at any time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intervention group will perform a therapeutic exercise program combined with RMT
  Interventions: Device: Therapeutic exercise program combined with RMT
- Control group (Sham Comparator): Control group will perform the same therapeutic exercise program combined with sham RMT
  Interventions: Device: Therapeutic exercise program combined with sham RMT

INTERVENTIONS:
Device: Therapeutic exercise program combined with RMT — For the RMT protocol, the Orygen-dual valve® device will be used. Each participant will start with a load of 30% of the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP). Once every 10 days, the performance will be reviewed and the resistance will be increased by 10cmH2O of the initial MIP/MEP of each patient. Each session will consist of breathing through the device for 20 minutes (10 minutes dedicated to each muscle group). This process will be repeated once a day, five days a week, for eight weeks.
  The therapeutic exercise program will be common to both groups and will be carried out at CHUAC hospital, in group sessions. The sessions will be held three days a week, for eight weeks. Each session will consist of a 10-minute warm-up part, 45 minutes of the main part (aerobic and strength-resistance exercise), and five minutes of cooling down.
  Arms: Intervention group
Device: Therapeutic exercise program combined with sham RMT — The sham RMT protocol will have the same frequency as in the intervention group. The therapeutic exercise program will be common to both groups and will be carried out at CHUAC hospital, in group sessions. The sessions will be held three days a week, for eight weeks. Each session will consist of a 10-minute warm-up part, 45 minutes of the main part (aerobic and strength-resistance exercise), and five minutes of cooling down.
  Arms: Control group

SUMMARY:
Stroke has a significant impact on morbidity, mortality and healthcare expenditure globally. In addition to the motor and cognitive consequences, as well as on functional independence and social participation, it can produce alterations in the respiratory function. Scientific evidence supports the application of both therapeutic exercise programs and respiratory muscle training (RMT). However, studies that combine both interventions are limited, and to date no study has been published that examines the effectiveness of this combination in the subacute phase of stroke, which is the one that presents the widest range of neuroplasticity. Objectives: To analyze the effects of a combined therapeutic exercise and RMT program, compared to the therapeutic exercise and sham RMT program, on different variables related to functional, respiratory, swallowing and speech/voice capacity, in patients in the subacute phase of a stroke. Type of research: double-blind randomized controlled clinical trial. Design: The study will be carried out at the University Hospital Complex of A Coruña (CHUAC), where 64 patients with more than three and less than six months of evolution after a stroke will be recruited. Participants will be randomly assigned to two groups: the intervention group will perform a combined therapeutic exercise and RMT program, while the control group will combine the same therapeutic exercise program and sham RMT. The duration of the intervention will be eight weeks. The therapeutic exercise program will be carried out three days per week and will consist of a cardiovascular exercise part and a strength-endurance part. The RMT protocol will involve both the inspiratory and expiratory muscles, using the Orygen-Dual Valve® device. The control group will use the same valve but without resistance, generating a sham RMT. It will have a frequency of five days per week and will be carried out at the home of each patient. Additionally, half the subjects in the intervention group will continue the RMT protocol once the eight-week period has ended, with a frequency of two days per week, until the six-month follow-up. Possible differences between groups will be analyzed before and after the intervention, and at three and six months of follow-up, in relation to the following domains: functional capacity, functional independence, lung and respiratory muscle function, swallowing and speech/voice function, respiratory signs and symptoms, and quality of life.

DETAILED DESCRIPTION:
This protocol is designed to analyze the effects of a therapeutic exercise program combined with an RMT protocol in patients with subacute stroke, compared to another group that will perform the therapeutic exercise program combined with sham RMT in relation to different functional variables.

Sample size assessment: The sample size calculation was performed using the G*Power software and based on the 6 Minute Walk Test (6MWT), chosen as the main variable. The minimum clinically important difference (MCID) data from the study by Fulk et al. (MCID=130) and the standard deviation (SD) from the study by Baker et al. (conducted in patients with subacute stroke in the United Kingdom, SD=143) were used. For a two-sided hypothesis, with a statistical power of 90% and a significance level of 0.05, a sample size of 32 subjects per group would be required (assuming a 20% loss over the course of the study). Additionally, a pilot phase will be developed at the beginning of the study with eight other subjects who will not be part of the final sample, in order study the feasibility of the project.

Plan for missing data: At the end of each assessment session, all questionnaires will be checked to ensure they are complete and filled out correctly. If a participant does not attend a session, they will be phone called and rescheduled for that session. In cases where data are reported as missing, unavailable, or uninterpretable due to inconsistencies or out-of-range results, a plan will be implemented to manage these cases. Strategies will include imputing missing data and excluding cases.

Statistical analysis plan: Anaconda® software and the Python 3.8.8 programming language will be used. A descriptive analysis of the variables included in the study will be performed initially. For qualitative variables, absolute frequencies and percentages will be presented, and for quantitative variables, measures of central tendency (mean/median) and dispersion (range/standard deviation) will be presented, depending on whether they are normal or non-normal. The normality of the sample will be tested using the Shapiro-Wilk test. Per-protocol and intention-to-treat analyses will be performed to determine the effectiveness of the treatment both under ideal conditions of protocol adherence and in a more realistic context of losses throughout the intervention. To compare the results of the outcome measures between the study groups throughout the intervention, a repeated-measures ANOVA will be applied with a within-subject factor, time, which has four levels (pre-training, post-training, and at three and six months post-training), and a between-subject factor, the type of intervention (therapeutic exercise + RMT or therapeutic exercise + sham RMT). Another repeated-measures ANOVA will be applied with the same within-subject factor, and the presence or absence of maintenance sessions as a between-subject factor (only for the intervention group). The level of statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria

* Those diagnosed with a first stroke occurring three to six months after the onset (subacute phase).
* Those aged 18 years or older.
* Those able to walk at least 10 meters, with or without walking aids and/or physical assistance from another person.

Exclusion Criteria:

* Those with recurrent stroke.
* Those with a history of chronic respiratory disease.
* Those with other underlying neurological diseases with impaired functionality prior to the stroke.
* Those with other cardiovascular or metabolic diseases in an unstable phase.
* Those with severe cognitive deficits that impede understanding of the assessment tests and/or the intervention.
* Those with severe facial paralysis that impedes proper performance of pulmonary function and respiratory muscle strength tests.
* Those with a prior participation in a RMT program.
* Those who participate in a cardiovascular and/or strength-endurance training program at the time of the study.
* Those with any of the contraindications to performing the tests included in the study protocol: spirometry, respiratory muscle strength and endurance tests, and 6MWT.
* Those with any of the contraindications to physical exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | The 6MWT will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The metric used to characterize the primary outcome measure will be the 6MWT. The 6MWT is a constant-load walking test that evaluates submaximal functional capacity. It consists of determining the distance a patient is able to walk at the maximum possible speed in six minutes, using standardized instructions. It will be carried out following the international standards of the American Thoracic Society (ATS) and the European Respiratory Society (ERS). The test will be performed in a hallway, with two markers delimiting the 30-meter distance. Every minute during the test, oxygen saturation, heart rate (HR), and dyspnea and fatigue of the lower limbs will be recorded, and blood pressure (BP) will be measured both before and after the test. In the first assessment session, two attempts will be made due to the learning effect, separated by a 30-minute rest period or as long as necessary until vital signs recover. A single attempt will be made in subsequent measurements.

SECONDARY OUTCOMES:
Sociodemographic data | The personal interview will take place once, before the intervention.
  Description: The following characteristics will be collected during the personal interview:(15,16)
  * Sociodemographic data: sex, age, nationality, employment status.
  * Toxic habits: information on smoking habits.
  * Medical history.
  * Medication use.
  * Information on the stroke: time elapsed, type, affected region.
  * Rehabilitation process: type, disciplines involved, weekly duration, technical aids.
Anthropometrics | Height, weight and BMI will be recorded in the first session (before intervention), and weight and BMI will be recorded in all assessment sessions (before and after intervention, and at the 3rd and 6th month of follow-up).
  Height, weight, and body mass index (BMI) will be recorded. Weight and height will be measured without shoes and without clothing that significantly increases weight and is easy to remove. Participants must also remove any items they may carry in their pockets that increase their weight (e.g., keys, cell phone, or wallet). BMI will be calculated using the formula BMI = weight (kg) / height (m2).
Upper and lower limb motor function | The MI will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  It will be assessed through the motricity index (MI). It is an ordinal method for measuring motor function and limb strength developed by Demeurisse et al. in 1980. It assesses the following movements: digital pinch between the thumb and index finger, elbow flexion, shoulder abduction, ankle dorsiflexion, knee extension, and hip flexion. It has a minimum score of 0 and a maximum of 100, with each test being given a value between 0 and 33. All tests are performed with the patient in a sitting position.
Fall risk | The TUG will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Timed Up and Go test (TUG) assesses mobility, balance, gait ability, and fall risk. The test begins with the patient seated in a chair with their back against the backrest. Upon command from the therapist, the patient must rise from the chair, walk three meters as quickly as possible to a marker (e.g., a cone), turn around the marker, return to the chair, and sit down. Timing begins upon the therapist's command to rise and ends when the patient is seated again. One attempt will be performed, accompanied by a practice pretest that will not be included in the score. For the stroke population, it has a minimum detectable change of 2.9 seconds and excellent test-retest reliability and criterion- and construct-related validity.
Balance | The BBS will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  It will be assessed using the Berg Balance Scale (BBS), which is an objective 14-item measure that evaluates static balance and the risk of falling in adults. The items that comprise it include static and dynamic activities of varying difficulty. The scores for each item range from 0 to 4, depending on the execution of the activity evaluated. Finally, the scores for all items are summed (maximum score = 56). The Berg scale has been frequently used in other studies with stroke samples, since it is associated with quality of life, and is sensitive (80%) and specific (78%) in identifying subjects at risk of falling after a stroke. In addition, it has excellent test-retest reliability, inter- and intra-rater reliability, internal consistency, criterion validity, and construct validity in the stroke population.
Lower limb strength | The 5TSTS will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Five Times Sit to Stand test (5TSTS) provides a method for quantifying functional lower extremity strength and identifying movement strategies that a patient uses to complete a transfer. The test begins with the patient sitting in a chair, arms crossed over the chest and back against the backrest. At the therapist's command, the patient must rise from the chair and return to sitting for five repetitions, as quickly as possible. Timing ends when the patient reaches the sitting position after the last repetition. An attempt will be made, accompanied by a pre-test practice that will not be included in the score. Failure to complete the five repetitions without assistance or use of the upper extremities indicates test failure. The test has a cutoff point of 12 seconds to discriminate between healthy subjects, the elderly, and those with chronic stroke.
Functional independence | The FIM will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Functional Independence Measure (FIM) provides a uniform system for measuring disability based on the International Classification of Functioning, Disability and Health (ICF). It measures a patient's level of disability and indicates the amount of assistance required to perform ADLs. Tasks are rated on a seven-point ordinal scale ranging from full assistance (or total dependence) to complete independence. Scores range from 18 (lowest) to 126 (highest), indicating the level of function. It contains 18 items, comprised of 13 motor tasks and five cognitive tasks. This scale has an MCID of 22 points in stroke subjects and exhibits excellent internal consistency and criterion validity, adequate construct validity, minimal ceiling and floor effects, and high sensitivity in stroke patients.
Functional ambulation | The FAC will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Functional Ambulation Category (FAC) assesses the patient's dependence for functional gait. The evaluator must check one of the following six boxes:
  0) The patient is unable to walk or requires assistance from two or more people.
  1. The patient requires firm, continuous support from a person to assist with weight bearing and balance.
  2. The patient requires continuous or intermittent support from a person to assist with balance and coordination.
  3. The patient requires verbal supervision or assistance from a person without physical contact.
  4. The patient can walk independently on level ground but requires assistance on stairs, slopes, or uneven surfaces.
  5. The patient can walk independently anywhere. A difference greater than four points in stroke patients has a sensitivity of 100% and a specificity of 78% in predicting community ambulation at six months. It also presents excellent test-retest reliability values and both intra-rater and inter-rater reliability.
Pulmonary function (FEV1/FVC) | The forced spirometry will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  Pulmonary volumes and flows will be obtained by forced spirometry, which consists of a maximum deep inspiration followed by a forced and sustained expiration through a spirometer. Additionally, another maximum inspiration will be performed at the end of the maneuver to obtain an inspiratory branch in the graph resulting from the test, as a quality criterion. The patient will remain seated during the test and will use a nose clip while executing the maneuvers. Forced spirometry will be performed following the recommendations of the ATS and ERS, and using a Datospir Aira spirometer (Sibelmed®, Barcelona, Spain). A minimum of three technically acceptable maneuvers will be obtained, with two being reproducible (<150 ml or <5% forced vital capacity (FVC) or forced expiratory volume in 1 second (FEV1) difference). FVC and FEV1 will be recorded. FVC and FEV1 will be combined to report FEV1/FVC.
Pulmonary function (PEF) | The forced spirometry will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  Pulmonary volumes and flows will be obtained by forced spirometry. Forced spirometry will be performed following the recommendations of the ATS and ERS, and using a Datospir Aira spirometer (Sibelmed®, Barcelona, Spain). Peak expiratory flow (PEF) will be obtained.
Pulmonary function (FEF25-75%) | The forced spirometry will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  Pulmonary volumes and flows will be obtained by forced spirometry. Forced spirometry will be performed following the recommendations of the ATS and ERS, and using a Datospir Aira spirometer (Sibelmed®, Barcelona, Spain). Forced expiratory flow between 25% and 75% of the FVC (FEF25-75%) will be obtained.
Strength of the inspiratory and expiratory muscles | The maximal respiratory pressures will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  Respiratory muscle strength will be obtained from the MEP and MIP. The recommendations of the Spanish Society of Pulmonology and Thoracic Surgery (SEPAR) will be followed. The measures will be determined using a pressure transducer with a diving-type mouthpiece, and the patient will perform the maneuvers in a sitting position with a nose clip. Forced and maximum expiration and inspiration will be performed, respectively, for three to five seconds, trying to maintain a constant force against the resistance offered by the device. The MicroRPM® Carefusion device (Vyaire Medical GmbH, Hoechberg, Germany) will be used, connected to the PUMA® software (Vyaire Medical GmbH, Hoechberg, Germany). A minimum of six maneuvers will be performed (out of a maximum of ten), with the goal of obtaining three technically correct, reproducible maneuvers with a variation of less than 5%.
Cough capacity | The PCF will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  It will be measured using a portable peak cough flow (PCF) meter connected to an orofacial mask (to prevent potential air leaks in the presence of mild facial paralysis), designed to quantify the maximum air flow expelled during a forced cough. This procedure evaluates the effectiveness of coughing in clearing secretions from the airways and is especially relevant in patients with neuromuscular or respiratory conditions. The patients will perform the maneuver in a seated position. They will be instructed to take a maximum inspiration from total lung capacity, after which they will adjust the orofacial mask around their mouth and cough forcefully. The device records the maximum air flow generated during the cough, expressed in liters per minute (L/min). Three attempts will be made, and the highest value will be recorded.
Severity of dysphagia | The GUSS will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Gugging Swallowing Screen (GUSS) is a bedside dysphagia screening tool for patients with acute stroke. It assesses the severity of dysphagia as well as the level of aspiration. It evaluates the ability to swallow saliva, semisolid, liquid, and solid textures. It also notes the presence of a cough or throat clearing at rest, as well as changes in voice. Oxygen saturation is monitored using a pulse oximeter during the test. Several studies have reported that the GUSS has a sensitivity of approximately 100% and a specificity of 50% to 69%.
Swallowing-related quality of life | The SWAL-QoL will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Swallowing Quality of Life Questionnaire (SWAL-QoL) is a self-administered questionnaire designed to assess quality of life in patients with oropharyngeal dysphagia. It consists of 44 items divided into 11 different domains. Each item is scored on a 5-point Likert scale. Each item is weighted and summed to obtain an overall score (0-100), with a lower score indicating poorer swallowing-related quality of life.
Voice parameters | The PRAAT recordings will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  Perceptual auditory assessment is the gold standard for defining voice disorders and providing an immediate measure of voice severity. PRAAT is a freely distributed program widely used in clinical practice. This program performs an acoustic analysis of the voice, providing objective information. It analyzes the average fundamental frequency, intensity, and all its variations. It provides disturbance indices and irregularity and noise measurements, which are used to analyze the harmonic component and emission regulation. The sample recording should be made at a frequency of 20,000 hertz (Hz), with ambient noise less than 50 decibels (dB), and the microphone should be placed at a distance of 10 centimeters, at an angle of 45° to 90°. Each patient is recorded saying a simple sentence at a comfortable pitch and intensity, recording three attempts to assess whether there is variability in vocal quality, one slightly more intense attempt to assess possible changes in quality.
Vocal quality | The GRABS scale will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The GRABS scale is the most reliable and widely used scale for the perceptual assessment of vocal quality. It consists of five parameters and four categories based on the severity of the disorder. These parameters are: G (grade), which assesses the overall degree of vocal disorder, dysphonia, or hoarseness; R (roughness), which assesses hoarseness and harshness; A (asthenic), which assesses the degree of asthenia and fatigue in the voice; B (breathy), which assesses a voice that is airy, muffled, or breathy; and S (strain), which assesses a tense, spastic, and constricted voice. Scores range from 0 to 3, with 0 being normal, 1 being mild, 2 being moderate, and 3 being severe. This scale has been validated and used in several studies and exhibits high diagnostic quality. It is a non-invasive test that is easy to use, requires no training for its application and does not require a high cost. The sample is collected through conversational speech heard during the interview.
Aerodynamics (MPT) | The aerodynamics will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  Maximum Phonation Time (MPT) consists of producing the vowel /a/ at a comfortable intensity and pitch for as long as possible. A prior demonstration is required. Three attempts are made, selecting the longest one to compare with the standard. If the value obtained is less than ten seconds, it would indicate abnormal respiratory function, poor glottal closure, or exaggerated glottal closure.
Aerodynamics (MBT) | The aerodynamics will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  Maximum blow time (MBT) allows the relationship between phonation and expiration to be analyzed through the so-called s/z ratio.
Aerodynamics (s/z ratio) | The aerodynamics will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The s/z ratio or phonorespiratory coefficient is the result of dividing the maximum emission time of a consonant /s/ by the maximum phonation time of an /a/, with the purpose of relating pulmonary and laryngeal function. Under normal circumstances, it should be approximately 1. When glottal efficiency is impaired, high values are obtained, with 1.4 being the normal limit.
Severity of dysarthria | The item 10 of the NIHSS will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The National Institute of Health Stroke Scale (NIHSS) will be used. This scale measures the severity of symptoms associated with a stroke, is used as a quantitative measure of neurological deficit and has good psychometric properties. Item 10, dedicated to dysarthria, will be recorded: a speech sample is obtained from the patient, asking them to read or repeat a series of words. It will be scored as follows: 0 = normal; 1 = mild to moderate dysarthria (can be understood with some difficulty); 2 = severe dysarthria (unintelligible or anarthria); 9 = unverifiable, if the patient is intubated or has other physical barriers to speech production (the justification for this choice must be given).
Dyspnea | The mMRC will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Modified Medical Research Council (mMRC) dyspnea scale determines the severity of shortness of breath during everyday activities, classified into 5 grades:
  0) No dyspnea, except with intense exercise.
  1. Dyspnea when walking briskly or climbing a gentle slope.
  2. Difficulty maintaining a pace when walking on level ground or keeping pace with other people of the same age.
  3. Need to stop after walking 100 meters or a few minutes.
  4. Severe dyspnea resulting in inability to leave the house or dress without assistance.
  This scale is recommended by various clinical practice guidelines and is used as an inclusion criterion for clinical trials.
Self-perceived effort | The Modified Borg Scale will be assessed before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Modified Borg Scale measures self-rated exertion, as determined by dyspnea and fatigue, during physical activity. It has the potential to provide rapid and easy information on a patient's subjective state of dyspnea and fatigue. It has 11 levels, from 0 (minimum) to 10 (maximum). It is a valid and reliable assessment tool for dyspnea.
Respiratory complications | The number and type of respiratory complications will be registered at baseline and until the 6-month follow-up period.
  They will be recorded through an interview and review of medical history. The following situations are understood to be respiratory complications: hospital admissions for respiratory reasons, emergency room visits for respiratory reasons, and/or lung infections requiring medication.
Quality of life (SIS-16) | The SIS-16 will be administered before the intervention, at the end of it (after 8 weeks) and at 3rd and 6th month of follow-up.
  The Stroke Impact Scale (SIS-16) assesses physical function after stroke. The SIS-16 consists of 16 items from the four physical domains (strength, hand function, mobility, and ADL/instrumental ADL) of the SIS 3.0. It has an MCID of 9.4-14.1 for subacute stroke and excellent test-retest reliability, internal consistency, and criterion- and construct-related validity.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lista Paz, PhD, Principal Investigator — Faculty of Physiotherapy, University of A Coruña.
Locations (1):
- University Hospital of A Coruña (CHUAC), A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data collected in this study, and in accordance with the data protection regulations of Spain and Europe, we are unable to share IPD. Our institutional and ethical guidelines prioritize participant confidentiality and privacy, ensuring that all data handling adheres to the highest standards of data protection.

REFERENCES:
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Fulk GD, Ludwig M, Dunning K, Golden S, Boyne P, West T. How much change in the stroke impact scale-16 is important to people who have experienced a stroke? Top Stroke Rehabil. 2010 Nov-Dec;17(6):477-83. doi: 10.1310/tsr1706-477. PMID 21239371
- [Background] Chou CY, Ou YC, Chiang TR. Psychometric comparisons of four disease-specific health-related quality of life measures for stroke survivors. Clin Rehabil. 2015 Aug;29(8):816-29. doi: 10.1177/0269215514555137. Epub 2014 Oct 28. PMID 25352615
- [Background] Duncan PW, Lai SM, Bode RK, Perera S, DeRosa J. Stroke Impact Scale-16: A brief assessment of physical function. Neurology. 2003 Jan 28;60(2):291-6. doi: 10.1212/01.wnl.0000041493.65665.d6. PMID 12552047
- [Background] Messaggi-Sartor M, Guillen-Sola A, Depolo M, Duarte E, Rodriguez DA, Barrera MC, Barreiro E, Escalada F, Orozco-Levi M, Marco E. Inspiratory and expiratory muscle training in subacute stroke: A randomized clinical trial. Neurology. 2015 Aug 18;85(7):564-72. doi: 10.1212/WNL.0000000000001827. Epub 2015 Jul 15. PMID 26180145
- [Background] Kendrick KR, Baxi SC, Smith RM. Usefulness of the modified 0-10 Borg scale in assessing the degree of dyspnea in patients with COPD and asthma. J Emerg Nurs. 2000 Jun;26(3):216-22. doi: 10.1016/s0099-1767(00)90093-x. PMID 10839848
- [Background] Sunjaya A, Poulos L, Reddel H, Jenkins C. Qualitative validation of the modified Medical Research Council (mMRC) dyspnoea scale as a patient-reported measure of breathlessness severity. Respir Med. 2022 Nov;203:106984. doi: 10.1016/j.rmed.2022.106984. Epub 2022 Sep 9. PMID 36179385
- [Background] Adams HP Jr, Davis PH, Leira EC, Chang KC, Bendixen BH, Clarke WR, Woolson RF, Hansen MD. Baseline NIH Stroke Scale score strongly predicts outcome after stroke: A report of the Trial of Org 10172 in Acute Stroke Treatment (TOAST). Neurology. 1999 Jul 13;53(1):126-31. doi: 10.1212/wnl.53.1.126. PMID 10408548
- [Background] Lee Y, Kim G, Kwon S. The Usefulness of Auditory Perceptual Assessment and Acoustic Analysis for Classifying the Voice Severity. J Voice. 2020 Nov;34(6):884-893. doi: 10.1016/j.jvoice.2019.04.013. Epub 2019 May 17. PMID 31104881
- [Background] Chandrashekaraiah B, N S, K PT. Impact of Effortful Swallow with Progressive Resistance on Swallow Safety, Efficiency and Quality of Life in Individuals with Post-Stroke Dysphagia: Analysis Using DIGEST- FEES and SWAL-QOL. Indian J Otolaryngol Head Neck Surg. 2023 Dec;75(4):2836-2841. doi: 10.1007/s12070-023-03846-7. Epub 2023 May 17. PMID 37974700
- [Background] Trapl M, Enderle P, Nowotny M, Teuschl Y, Matz K, Dachenhausen A, Brainin M. Dysphagia bedside screening for acute-stroke patients: the Gugging Swallowing Screen. Stroke. 2007 Nov;38(11):2948-52. doi: 10.1161/STROKEAHA.107.483933. Epub 2007 Sep 20. PMID 17885261
- [Background] Bhakta NR, McGowan A, Ramsey KA, Borg B, Kivastik J, Knight SL, Sylvester K, Burgos F, Swenson ER, McCarthy K, Cooper BG, Garcia-Rio F, Skloot G, McCormack M, Mottram C, Irvin CG, Steenbruggen I, Coates AL, Kaminsky DA. European Respiratory Society/American Thoracic Society technical statement: standardisation of the measurement of lung volumes, 2023 update. Eur Respir J. 2023 Oct 12;62(4):2201519. doi: 10.1183/13993003.01519-2022. Print 2023 Oct. PMID 37500112
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Kollen B, Kwakkel G, Lindeman E. Time dependency of walking classification in stroke. Phys Ther. 2006 May;86(5):618-25. PMID 16649886
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Mehrholz J, Pohl M, Kugler J, Elsner B. The Improvement of Walking Ability Following Stroke. Dtsch Arztebl Int. 2018 Sep 28;115(39):639-645. doi: 10.3238/arztebl.2018.0639. PMID 30375325
- [Background] Ward I, Pivko S, Brooks G, Parkin K. Validity of the stroke rehabilitation assessment of movement scale in acute rehabilitation: a comparison with the functional independence measure and stroke impact scale-16. PM R. 2011 Nov;3(11):1013-21. doi: 10.1016/j.pmrj.2011.08.537. PMID 22108228
- [Background] Salter K, Jutai J, Foley N, Teasell R. Clinical Outcome Variables Scale: A retrospective validation study in patients after stroke. J Rehabil Med. 2010 Jul;42(7):609-13. doi: 10.2340/16501977-0567. PMID 20603689
- [Background] Inouye M, Hashimoto H, Mio T, Sumino K. Influence of admission functional status on functional change after stroke rehabilitation. Am J Phys Med Rehabil. 2001 Feb;80(2):121-5; quiz 126, 146. doi: 10.1097/00002060-200102000-00008. PMID 11212012
- [Background] Hsueh IP, Lin JH, Jeng JS, Hsieh CL. Comparison of the psychometric characteristics of the functional independence measure, 5 item Barthel index, and 10 item Barthel index in patients with stroke. J Neurol Neurosurg Psychiatry. 2002 Aug;73(2):188-90. doi: 10.1136/jnnp.73.2.188. PMID 12122181
- [Background] Denti L, Agosti M, Franceschini M. Outcome predictors of rehabilitation for first stroke in the elderly. Eur J Phys Rehabil Med. 2008 Mar;44(1):3-11. PMID 18385622
- [Background] Brock KA, Goldie PA, Greenwood KM. Evaluating the effectiveness of stroke rehabilitation: choosing a discriminative measure. Arch Phys Med Rehabil. 2002 Jan;83(1):92-9. doi: 10.1053/apmr.2002.27348. PMID 11782838
- [Background] Beninato M, Gill-Body KM, Salles S, Stark PC, Black-Schaffer RM, Stein J. Determination of the minimal clinically important difference in the FIM instrument in patients with stroke. Arch Phys Med Rehabil. 2006 Jan;87(1):32-9. doi: 10.1016/j.apmr.2005.08.130. PMID 16401435
- [Background] Mong Y, Teo TW, Ng SS. 5-repetition sit-to-stand test in subjects with chronic stroke: reliability and validity. Arch Phys Med Rehabil. 2010 Mar;91(3):407-13. doi: 10.1016/j.apmr.2009.10.030. PMID 20298832
- [Background] Beninato M, Portney LG, Sullivan PE. Using the International Classification of Functioning, Disability and Health as a framework to examine the association between falls and clinical assessment tools in people with stroke. Phys Ther. 2009 Aug;89(8):816-25. doi: 10.2522/ptj.20080160. Epub 2009 Jun 11. PMID 19520733
- [Background] Wee JY, Wong H, Palepu A. Validation of the Berg Balance Scale as a predictor of length of stay and discharge destination in stroke rehabilitation. Arch Phys Med Rehabil. 2003 May;84(5):731-5. doi: 10.1016/s0003-9993(02)04940-7. PMID 12736890
- [Background] Alghadir AH, Al-Eisa ES, Anwer S, Sarkar B. Reliability, validity, and responsiveness of three scales for measuring balance in patients with chronic stroke. BMC Neurol. 2018 Sep 13;18(1):141. doi: 10.1186/s12883-018-1146-9. PMID 30213258
- [Background] Knorr S, Brouwer B, Garland SJ. Validity of the Community Balance and Mobility Scale in community-dwelling persons after stroke. Arch Phys Med Rehabil. 2010 Jun;91(6):890-6. doi: 10.1016/j.apmr.2010.02.010. PMID 20510980
- [Background] Flansbjer UB, Holmback AM, Downham D, Patten C, Lexell J. Reliability of gait performance tests in men and women with hemiparesis after stroke. J Rehabil Med. 2005 Mar;37(2):75-82. doi: 10.1080/16501970410017215. PMID 15788341
- [Background] Andersson AG, Kamwendo K, Seiger A, Appelros P. How to identify potential fallers in a stroke unit: validity indexes of 4 test methods. J Rehabil Med. 2006 May;38(3):186-91. doi: 10.1080/16501970500478023. PMID 16702086
- [Background] Collin C, Wade D. Assessing motor impairment after stroke: a pilot reliability study. J Neurol Neurosurg Psychiatry. 1990 Jul;53(7):576-9. doi: 10.1136/jnnp.53.7.576. PMID 2391521
- [Background] Thilarajah S, Mentiplay BF, Bower KJ, Tan D, Pua YH, Williams G, Koh G, Clark RA. Factors Associated With Post-Stroke Physical Activity: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Sep;99(9):1876-1889. doi: 10.1016/j.apmr.2017.09.117. Epub 2017 Oct 19. PMID 29056502
- [Background] Lee J, Stone AJ. Combined Aerobic and Resistance Training for Cardiorespiratory Fitness, Muscle Strength, and Walking Capacity after Stroke: A Systematic Review and Meta-Analysis. J Stroke Cerebrovasc Dis. 2020 Jan;29(1):104498. doi: 10.1016/j.jstrokecerebrovasdis.2019.104498. Epub 2019 Nov 13. PMID 31732460
- [Background] Fulk GD, Echternach JL, Nof L, O'Sullivan S. Clinometric properties of the six-minute walk test in individuals undergoing rehabilitation poststroke. Physiother Theory Pract. 2008 May-Jun;24(3):195-204. doi: 10.1080/09593980701588284. PMID 18569856
- [Background] Macchiavelli A, Giffone A, Ferrarello F, Paci M. Reliability of the six-minute walk test in individuals with stroke: systematic review and meta-analysis. Neurol Sci. 2021 Jan;42(1):81-87. doi: 10.1007/s10072-020-04829-0. Epub 2020 Oct 16. PMID 33064231
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Hendrey G, Holland AE, Mentiplay BF, Clark RA, Williams G. Do Trials of Resistance Training to Improve Mobility After Stroke Adhere to the American College of Sports Medicine Guidelines? A Systematic Review. Arch Phys Med Rehabil. 2018 Mar;99(3):584-597.e13. doi: 10.1016/j.apmr.2017.06.021. Epub 2017 Jul 26. PMID 28756248
- [Background] Eng JJ. Fitness and Mobility Exercise (FAME) Program for stroke. Top Geriatr Rehabil. 2010;26(4):310-323. doi: 10.1097/TGR.0b013e3181fee736. PMID 22287825
- [Background] MacKay-Lyons M, Billinger SA, Eng JJ, Dromerick A, Giacomantonio N, Hafer-Macko C, Macko R, Nguyen E, Prior P, Suskin N, Tang A, Thornton M, Unsworth K. Aerobic Exercise Recommendations to Optimize Best Practices in Care After Stroke: AEROBICS 2019 Update. Phys Ther. 2020 Jan 23;100(1):149-156. doi: 10.1093/ptj/pzz153. PMID 31596465
- [Background] Sutbeyaz ST, Koseoglu F, Inan L, Coskun O. Respiratory muscle training improves cardiopulmonary function and exercise tolerance in subjects with subacute stroke: a randomized controlled trial. Clin Rehabil. 2010 Mar;24(3):240-50. doi: 10.1177/0269215509358932. Epub 2010 Feb 15. PMID 20156979
- [Background] Lista-Paz A, Langer D, Barral-Fernandez M, Quintela-Del-Rio A, Gimeno-Santos E, Arbillaga-Etxarri A, Torres-Castro R, Vilaro Casamitjana J, Varas de la Fuente AB, Serrano Veguillas C, Bravo Cortes P, Martin Cortijo C, Garcia Delgado E, Herrero-Cortina B, Valera JL, Fregonezi GAF, Gonzalez Montanez C, Martin-Valero R, Francin-Gallego M, Sanesteban Hermida Y, Gimenez Moolhuyzen E, Alvarez Rivas J, Rios-Cortes AT, Souto-Camba S, Gonzalez-Doniz L. Maximal Respiratory Pressure Reference Equations in Healthy Adults and Cut-off Points for Defining Respiratory Muscle Weakness. Arch Bronconeumol. 2023 Dec;59(12):813-820. doi: 10.1016/j.arbres.2023.08.016. Epub 2023 Sep 29. English, Spanish. PMID 37839949
- [Background] Parreiras de Menezes KK, Nascimento LR, Ada L, Avelino PR, Polese JC, Mota Alvarenga MT, Barbosa MH, Teixeira-Salmela LF. High-Intensity Respiratory Muscle Training Improves Strength and Dyspnea Poststroke: A Double-Blind Randomized Trial. Arch Phys Med Rehabil. 2019 Feb;100(2):205-212. doi: 10.1016/j.apmr.2018.09.115. Epub 2018 Oct 12. PMID 30316960
- [Background] Gomes-Neto M, Saquetto MB, Silva CM, Carvalho VO, Ribeiro N, Conceicao CS. Effects of Respiratory Muscle Training on Respiratory Function, Respiratory Muscle Strength, and Exercise Tolerance in Patients Poststroke: A Systematic Review With Meta-Analysis. Arch Phys Med Rehabil. 2016 Nov;97(11):1994-2001. doi: 10.1016/j.apmr.2016.04.018. Epub 2016 May 20. PMID 27216224
- [Background] Fabero-Garrido R, Del Corral T, Angulo-Diaz-Parreno S, Plaza-Manzano G, Martin-Casas P, Cleland JA, Fernandez-de-Las-Penas C, Lopez-de-Uralde-Villanueva I. Respiratory muscle training improves exercise tolerance and respiratory muscle function/structure post-stroke at short term: A systematic review and meta-analysis. Ann Phys Rehabil Med. 2022 Sep;65(5):101596. doi: 10.1016/j.rehab.2021.101596. Epub 2021 Nov 18. PMID 34687960
- [Background] Clague-Baker N, Robinson T, Hagenberg A, Drewry S, Gillies C, Singh S. The validity and reliability of the Incremental Shuttle Walk Test and Six-minute Walk Test compared to an Incremental Cycle Test for people who have had a mild-to-moderate stroke. Physiotherapy. 2019 Jun;105(2):275-282. doi: 10.1016/j.physio.2018.12.005. Epub 2018 Dec 21. PMID 30954276
- [Background] Fulk GD, He Y. Minimal Clinically Important Difference of the 6-Minute Walk Test in People With Stroke. J Neurol Phys Ther. 2018 Oct;42(4):235-240. doi: 10.1097/NPT.0000000000000236. PMID 30138230